CLINICAL TRIAL: NCT05352789
Title: Exploration of Nutrition and Metabolic Prehabilitation Practices for Haematopoietic Stem Cell Transplant (HSCT) in UK and ROI Transplant Centres: A BSBMT Multi-centre Survey
Brief Title: Nutrition and Metabolic Prehabilitation in HSCT Patients UK and ROI. BSBMT Multi-centre Survey.
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other); University of Sheffield (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IDBSBMT
Record Dates: First submitted 2021-03-24; First posted 2022-04-29 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Haematological Malignancy; Bone Marrow Transplant Complications; Stem Cell Transplant Complications; Nutrition Aspect of Cancer; Nutritional and Metabolic Disease; Exercise Interventions; Prehabilitation
Keywords: nutrition; metabolism; exercise; bone marrow transplant; stem cell transplant; autologous transplant; allogeneic transplant; prehabilitation
MeSH Terms: conditions — Hematologic Neoplasms; Metabolic Diseases; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non validated Survey — Overall inclusion of metabolic and nutritional parameters in prehabilitation practices will be assessed as the proportion of each parameter conducted from the mandatory queries presents as yes/no/unsure responses for each centre. Intervention or process details for included parameters will be described based on the response variable. The survey presents 4 question formats; free text (thematic qualitative analysis), 5 and 6 point likert scales (proportional response), categorical data (proportional response) and yes/no/unsure response sets (Binary response (no and unsure - grouped). All categorical data versions are parameter dependent and response variables can be requested from the research team.

SUMMARY:
To explore current practices of nutrition and metabolic screening, assessment and management prior to Haematopoietic Stem Cell Transplant (HSCT) in UK and ROI transplant centres.

Nutrition and metabolic parameters assessed in the survey include glycaemic control, lipid function, liver function, nutritional screening, nutritional assessment, nutrition intervention (tube feeding, diet, micronutrient) and exercise.

This work will be used to inform the design of a UK dual centre feasibility study of personalised nutrition and metabolic care for HSCT patients prior to transplantation.

ELIGIBILITY:
Inclusion Criteria:

* BSBMT registered adult HSCT centres (including TYA services where patients have opted to be treated in an adult service pathways)
* Centres delivering either autologous or allogeneic stem cell transplants

Exclusion Criteria:

* All paediatric HSCT services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care professionals working within an adult HSCT setting
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
To understand the routine screening, assessment and management practices of nutritional and metabolic parameters prior to haematopoeitic stem cell transplantation in UK centres | Aug 20- March22
  full survey completion: see parameters below
Differences in frequency of glycaemic screening prior to HSCT across UK and ROI HSCT centres and between health professionals | Aug 20-March22
  a) Glycaemic screening will be assessed by 2 responses: How often would you measure blood glucose and urinary glucose prior to HSCT? (likert scale - Always, often, sometimes, rarely, never)
Differences in frequency of assessments of lipid profile screening prior to HSCT across UK and ROI HSCT centres and between health professionals | Aug 20-March22
  b. Lipid parameters: How often would you measure blood glucose and urinary glucose prior to HSCT? (likert scale - Always, often, sometimes, rarely, never)
Differences in frequency of assessments of liver and renal function prior to HSCT across UK and ROI HSCT centres and between health professionals | Aug 20-March22
  c. Liver and renal function screening frequency will be asked: 1. How often would you measure liver/kidney function as blood samples prior to HSCT? (likert scale - Always, often, sometimes, rarely, never); 2. How often would you measure liver/kidney function using a scan prior to HSCT? (likert scale - Always, often, sometimes, rarely, never)
Differences in nutritional screening and assessment practices done prior to HSCT across UK and ROI HSCT centres and between health professionals | Aug 20-March22
  d. Nutritional screening and assessment: Routine inclusion of nutritional screening and assessment practices prior to HSCT will be assessed using 4 mandatory questions, 3 - yes/no/unsure and 1 categorical question. Practical details of strategies of assessment and measurement will be assessed using 5 categorical questions and 6 free text questions.
Differences in body composition assessments given prior to HSCT across UK and ROI HSCT centres and between health professionals | Aug 20-March22
  e. Assessment of body composition: Routine inclusion of body composition assessment prior to HSCT will be assessed using 2 mandatory questions, 1 - yes/no/unsure and 1 categorical question. Practical details of strategies of assessment and measurement will be assessed using 2 categorical questions and 3 free text questions.
Differences in dietary advice given prior to HSCT across UK and ROI HSCT centres and between health professionals | Aug 20-March22
  f. Dietary advice: Routine inclusion of dietary advice prior to HSCT will be assessed using 3 mandatory questions, 1 - yes/no/unsure and 2 - five point likert scales (definitely = 4, very probably = 3, probably=2, probably not = 1, definitely not =0). Practical details of types of dietary advice and strategies for implementation will be assessed using 2 categorical questions, 2 free text questions and 3 - six point likert scaled consensus statements (Always= 5, very frequently = 4, occasionally = 3, rarely = 2, very rarely = 1, never = 0)
Differences in enteral feeding practices prior to HSCT across UK and ROI HSCT centres and between health professionals | Aug 20-March22
  g. Enteral feeding: Routine inclusion of enteral feeding prior to HSCT will be assessed using 2 mandatory questions, 1 - categorical. Practical details of types of enteral feeding tubes 2 questions (1 - categorical questions, 1 free text)
Differences in specialist dietary advice given prior to HSCT across UK and ROI HSCT centres and between health professionals | Aug 20-March22
  h. Micronutrient supplementation: Routine inclusion of micronutrient advice prior to HSCT will be assessed using 1 mandatory question, yes/no/unsure format. Practical details of micronutrient supplementation practices using 1 categorical questions and 1 free text question.
Differences in physical assessment, advice and delivery prior to HSCT across UK and ROI HSCT centres and between health professionals | Aug 20-March22
  i. Exercise: As part of routine practice how often do patients receive exercise advice prior to HSCT? (likert response: Always, often, sometimes, rarely, never); As part of "routine practice" how often do your patients have their activity levels measured prior to HSCT i.e. questionnaire or physical assessment? response: Always, often, sometimes, rarely, never); and 2 multi select questions to determine professionals delivering care.

SECONDARY OUTCOMES:
To understand perceptions on the role and value of prehabilitation in HSCT | Aug 20-March22
  a. Point of effectiveness: using responses from three questions; Do you think prehabilitation should be considered as part of future services for HSCT? (Yes/no/unsure); When in the HSCT pathway do you think a prehabilitation service could be introduced? Assessed via categorical data (Prior to diagnosis, at diagnosis prior to chemotherapy, during induction chemotherapy, end of induction chemotherapy, maintenance chemo, during HSCT assessment clinic, other than listed); Do you think any changes are needed to the Silver et al (2013) prehabilitation definition in order for it to be relevant to HSCT?* (yes/no/unsure); 2 x free text answers for concerns and barriers to implementation.
Perceptions on best composition of prehabilitation programme prior to HSCT. | Aug 20-March22
  a) This would be answered with two questions: How important do you think exercise, nutrition and psychological care are in prehabilitation programme for HSCT? (very important, important, moderately important, slightly important, not important) ; Are there any other components that you think should be considered as part of a prehabilitation programme for HSCT? (free text)
Description of current HSCT prehabilitation services in adult services in UK and ROI | Aug 20-March22
  2 x single select; What components of prehabilitation does your service include? (nutrition, psychology, exercise, other); Do you have a dedicated prehabilitation service for HSCT at your unit? (yes/no/unsure); Which other components are included as part of your prehabilitation programme for HSCT?

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom